CLINICAL TRIAL: NCT07051525
Title: Early Versus Late Stopping of Antibiotics in Adults With High Risk Haematological Malignancies/Receiving Cellular Therapies and Fever (ELSA- Adult)
Brief Title: Early Versus Late Stopping of Antibiotics in Adults With High-risk Hematological Malignancies/Receiving Cellular Therapies and Fever
Acronym: ELSA-Adult
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24/236; 2024.406 (Other: Royal Melbourne Hospital Research Office); ERM113654 (Other: Peter MacCallum Cancer Centre)
Record Dates: First submitted 2025-04-21; First posted 2025-07-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Leukemia; CART Therapy; Transplantation, Stem Cell; Infections, Bacterial
Keywords: EPIC; ELSA; Febrile neutropaenia; Febrile neutropenia; antibitoics
MeSH Terms: conditions — Leukemia; Bacterial Infections; Febrile Neutropenia

STUDY DESIGN:
Intervention Model Description: Intervention: Early discontinuation of empiric antibiotic therapy: ceasing antibiotics upon meeting all inclusion and no exclusion criteria Control: Standard of care: Continuing empiric antibiotics beyond resolution of fever for at least 96 hours and otherwise as per clinician's discretion (typically recovery of absolute neutrophil count (ANC) to >200 cells/mm3)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STOP - early discontinuation of empiric antibiotic therapy (Experimental): Short course antibiotics (STOP): Antibiotics will be commenced at onset of fever and stopped once afebrile for 48-96 hours and clinically stable.
  Interventions: Drug: Early antibiotic cessation alert
- SOC - standard of care continuation of empiric antibiotic therapy (No Intervention): Standard of care (SOC): Antibiotics will be commenced at onset of fever and continued for a duration as per clinician's discretion, typically until resolution of fever, clinical recovery and ANC ≥200- 500 cells/mm3.

INTERVENTIONS:
Drug: Early antibiotic cessation alert — For all patients, antibiotics will be commenced at onset of fever. For those in the intervention arm an alert will fire in the electronic medical record once a patient is afebrile for 48-96 hours and clinically stable.
  Arms: STOP - early discontinuation of empiric antibiotic therapy

SUMMARY:
Pre-neutropenic fever (PNF) (fever following chemotherapy but before developing low white cells) and neutropenic fever (NF) (fever in the setting of low white cells) are very common after chemotherapy for acute leukemia, bone marrow transplantation or Chimeric Antigen Receptor T-cell (CAR T) therapy. Often, there is no bacterial cause for fever found, and in the setting of a well patient with resolved fever, some studies have shown it to be safe to cease antibiotic therapy which was commenced at the onset of fever. This reduces the overall exposure to antibiotics, which can be beneficial to the patient (reduced risk of resistant bugs emerging, reduced serious side effects). However, some subgroups of high-risk patients have been underrepresented in these studies (in particular, those who have received a bone marrow transplant from a donor, those with longer duration of low white cells) and none have been performed in Australia, hence applying this data to our setting and patient groups is indirect and further data are needed. This study plans to recruit participants who have received chemotherapy for acute leukemia or a stem cell transplant (either their own cells or a donor's cells) or CAR T-cell therapy and perform a trial to compare early stopping of antibiotics (STOP arm) to the standard of care, which traditionally involves continuing antibiotics until the white cell count reaches above a specific threshold. The primary study outcome is duration of days free of antibiotics within 28 days of study allocation. The investigators will also observe for important clinical outcomes including rates of fever recurrence, bloodstream and other infections, intensive care admission and mortality. Patients will stay in hospital during this period, even in the setting of stopping antibiotics, and these antibiotics can be recommenced urgently according to the sepsis protocol if there is concern for infection.

DETAILED DESCRIPTION:
This study is designed to assess the safety, benefits and impacts of early cessation of empiric antibiotics in all fever (both pre-neutropenic (PNF) and neutropenic (NF)) that develops post conditioning or chemotherapy until count recovery in high-risk hematology patients who meet clear inclusion criteria. This is in recognition of the fact that both PNF and NF are often not infective in nature, and that cessation is likely an important and safe approach in both scenarios. Secondly, the patient's pre-neutropenic and neutropenic status is highly fluid and can rapidly change from one to the other (within a day), making strict definitions of neutropenia arbitrary and not particularly useful for implementation in the clinical setting. Furthermore, as a programmatic-type intervention that is embedded in clinical workflow, approaching high-risk patients with fever in a standardized way would enable consistency and inform clear and concise management protocols. Stratification will allow for assessment of each patient sub-group to provide more granular data.

As an Australian first, this study will exploit the full potential of electronic medical record (EMR) systems, embedding all key aspects of the trial including screening, randomization and data collection into standard clinical and EMR workflows. This highly novel and innovative clinical trial methodology has the potential to improve trial efficiency, data quality and transferability between healthcare centers and will systematically evaluate the barriers and enablers of embedded trials (ELSA-EMR).

The study hypothesizes that early cessation of antibiotics in adult patients with high risk fever is safe, acceptable, cost-effective and will minimize an unnecessarily prolonged health care intervention

ELIGIBILITY:
Inclusion Criteria:

Adult patients ( ≥18 years) who are receiving either:

* Conditioning chemotherapy for an autologous or allogeneic haematopoietic cell transplant or CAR T cell therapy, OR
* Induction remission chemotherapy for acute leukaemia,

AND develop fever ( ≥38degC) between time of initiation of chemotherapy/conditioning administration and ANC recovery to ≥500 cells/mm3 post the ANC nadir,

AND fever subsequently has settled (<38degC) for ≥48 and <96h hours.

[participants will be stratified into pre-neutropenic (ANC ≥500 cells/mm3) and neutropenic (ANC<500 cells/mm3) strata based on ANC level at 48 hours post fever onset, as per international consensus definition of neutropenic fever]

Exclusion Criteria:

* - Prolonged fever prior to defervescence (documented daily temperature ≥38.0°C for ≥ 5 days)
* Documented positive blood culture for bacteria since onset of fever episode and prior to randomisation
* Documented other infection (clinically or microbiologically defined) requiring antibacterial treatment
* Grade 2 or higher mucositis (WHO) or neutropenic enterocolitis
* Clinically unstable and/or admission to ICU at time of potential randomization
* Within 28 days of last randomization
* Prior randomization during current chemotherapy/conditioning cycle
* Pregnant or breastfeeding
* Currently being treated for CRS Grade 3 or 4, and/or ICANS Grade 3 or 4 (defined as per ASTCT Consensus Guidelines, Lee et al)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2027-12-05 (Estimated); Study Completion 2028-02-05 (Estimated)

PRIMARY OUTCOMES:
Days free of antibiotic therapy in 28 days post randomization (termed empiric antibiotic free days (EAFDs)) | 28 days after randomization
  The primary study outcome is duration of days free of antibiotics within 28 days of study allocation. Measured as antibiotic free days in last 28 days post fever onset

SECONDARY OUTCOMES:
Days alive and free of antibiotic therapy in 28 days post randomization | 28 days after randomization
  Days alive and free of antibiotic therapy in 28 days post randomization
Recurrence of fever (>38deg Celsius) beyond randomization | same episode of neutropenia - until ANC>500 cells/mm3
  Recurrence of fever (>38deg Celsius, confirmed on second reading within 1 hour) post randomization during the same episode of neutropenia, not associated with blood product transfusion
  * In CAR T treated patients, grade of cytokine release syndrome (CRS), immune-cell associated neurotoxicity (ICANS) at time of fever and any recurrent fever.
Number of occasions antibiotic therapy is recommenced with treatment intent | Within 28 days after randomization
  Number of events antibiotic therapy is recommenced with treatment intent (excluding prophylaxis)
Days of antibiotic therapy during neutropenic period | Neutropenic period - until ANC>500 cells/mm3
  Days of antibiotic therapy during neutropenic period until ANC>500 cells/mm3
Number of intensive care unit (ICU) admissions | pre-neutropenic and neutropenic period post randomization (until ANC>500 cells/mm3)
  Admission to intensive care for organ support during the same pre-neutropenic and neutropenic period post randomization
Number of events of clinical instability | 28 days after randomization
  Number of events of clinical instability (defined by blood pressure, oxygen saturations, respiratory rate and heart rate meeting at least 1 Medical Emergency Team (MET) call criteria or 2 clinical review criteria)
Number of events of new positive blood culture | 28 days after randomization
  Number of events of new positive blood culture post randomization (defined by CDC criteria)
28 day all-cause mortality and infection-related mortality | 28 days after randomization
  28 day all-cause mortality and infection-related mortality (as assessed by an independent data safety monitoring board)
Measure number of patient days of total hospital admission | Measure number of days of total hospital length of stay during enrolment (admission until discharge from hospital inpatient and HITH)
  Duration of in-hospital length of stay calculated from randomization date and time to discharge from hospital ward or Hospital-In-The-Home (HITH)
Total number of days of in-hospital length of stay | Total number of days of in-hospital length of stay
  Duration of in-hospital length of stay calculated from randomization date and time to discharge/transfer from in- hospital ward
Total hospital length of stay post randomisation | Total hospital length of stay post randomization to discharge (from ward or HITH)
  Duration of in-hospital length of stay calculated from randomization date and time to discharge from hospital ward or HITH
Number of unplanned hospital readmissions | within 60 days of randomization
  Unplanned readmission to hospital within 60 days of randomization, defined as any admission that is not due to planned chemotherapy, conditioning or routine neutropenic monitoring as per standard protocols.
Number of positive C.difficile infections | within 6 months of randomization
  Number of development of C.difficile infection (defined by diarrhea, positive toxin polymerase chain reaction (PCR) and lack of other cause) within 6 months of randomization
Number of antibiotic resistant infection or colonizations | within 180 days post randomization
  New antibiotic resistant (Methicillin-resistant Staphylococcus aureus (MRSA), Extended-Spectrum Beta-Lactamases (ESBL) producing Enterobacterales, Carbapenem-resistant Enterobacterales (CRE), Vancomycin-resistant Enterococcus (VRE) infection or colonization detected within 180 days post randomization
Number of Clinically defined infections during pre-neutropenic and neutropenic period | pre-neutropenic and neutropenic period until ANC>500 cells/mm3
  Number of Clinically defined infections during pre-neutropenic and neutropenic period
Number of clinically defined infections post randomization | post randomization until 28days
  Number of clinically defined infections post randomization
Number of microbiologically defined infections during pre-neutropenic and neutropenic period | during pre-neutropenic and neutropenic period until ANC>500 cells/mm3
  Number of microbiologically defined infections during pre-neutropenic and neutropenic period
Number of microbiologically defined infections post randomization | post randomization until 28days
  Number of microbiologically defined infections post randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Abby P Douglas, MBBS PhD FRACP, Principal Investigator — Peter MacCallum Cancer Centre; National Centre for Infections in Cancer
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No